CLINICAL TRIAL: NCT03300544
Title: A Phase I Study of Talimogene Laherparepvec (Talimogene Laherparepvec) With Neoadjuvant Chemotherapy and Radiation in Adenocarcinoma of the Rectum
Brief Title: Talimogene Laherparepvec, Chemotherapy, and Radiation Therapy Before Surgery in Treating Patients With Locally Advanced or Metastatic Rectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01844; NCI-2016-01844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10058; 10058 (Other: University of Texas MD Anderson Cancer Center LAO); 10058 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-03 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Rectal Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Rectal Adenocarcinoma; Stage III Rectal Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7; Stage IV Rectal Cancer AJCC v7; Stage IVA Rectal Cancer AJCC v7; Stage IVB Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Radiotherapy; Radiation; talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (T-VEC, capecitabine, chemoradiation) (Experimental): Patients receive talimogene laherparepvec intralesionally via endoscopy on weeks 1, 4, 6, and 8. Patients receive 5-fluorouracil IV by bolus and over 46 hours, leucovorin IV bolus, and oxaliplatin IV over 2 hours on weeks 2 and 4. Patients also receive capecitabine orally PO BID followed by radiation therapy for 28 fractions on days 1-5 of weeks 8-13. Patients undergo resection surgery on weeks 21-25.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Radiation: Radiation Therapy; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Radiation: Radiation Therapy — Undergo chemoradiation
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Talimogene Laherparepvec — Given intralesionally
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase I trial studies the best dose and side effects of talimogene laherparepvec in combination with 5-fluorouracil, leucovorin, oxaliplatin, capecitabine, and chemoradiation before surgery in treating patients with rectal cancer that has spread from where it started to nearby tissue and lymph nodes. Drugs used in immunotherapy, such as talimogene laherparepvec, may stimulate the body's immune system to fight tumor cells. Drugs used in chemotherapy, such as 5-fluorouracil, leucovorin, oxaliplatin, and capecitabine work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving talimogene laherparepvec, 5-fluorouracil, leucovorin, oxaliplatin, and capecitabine and chemoradiation before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the dose limiting toxicities (DLTs) and maximum tolerated dose (MTD) of talimogene laherparepvec in combination with chemotherapy and radiation in rectal cancer.

SECONDARY OBJECTIVES:

I. To establish safety and feasibility of the combination. II. To determine the neoadjuvant rectal (NAR) score of talimogene laherparepvec with chemotherapy and radiation.

EXPLORATORY OBJECTIVES:

I. To correlate genomic information including RAS, RAF mutation status with response, disease free survival (DFS) and/or overall survival (OS).

II. To determine immunomodulatory changes following talimogene laherparepvec, chemotherapy and radiation treatment including proportions of immune cell infiltrates in serially collected peripheral blood and/or frozen tumor samples (pre-, on treatment, and at post progression).

III. To identify magnetic resonance imaging (MRI)-based features including MRI circumferential margin (mrCRM) at baseline or post-therapy mrCRM, MRI tumor regression grade (mrTRG) to define determinants of response, DFS and OS.

IV. To determine the disease free survival (DFS) and overall survival (OS) of talimogene laherparepvec with chemotherapy and radiation in patients undergoing curative resection.

V. To determine the pathological complete response (pCR) rate of talimogene laherparepvec with chemotherapy and radiation.

OUTLINE: This is a dose-escalation study of talimogene laherparepvec.

Patients receive talimogene laherparepvec intralesionally via endoscopy on weeks 1, 4, 6, and 8. Patients receive 5-fluorouracil intravenously (IV) by bolus and over 46 hours, leucovorin IV bolus, and oxaliplatin IV over 2 hours on weeks 2 and 4. Patients also receive capecitabine orally (PO) twice daily (BID) followed by radiation therapy for 28 fractions on days 1-5 of weeks 8-13. Patients undergo resection surgery on weeks 21-25.

After completion of study treatment, patients are followed up for 30 days and up to 5 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation: Patients must have A) histologically or cytologically confirmed low lying (up to 6 cm of anal verge) rectal adenocarcinoma eligible for radiation therapy to rectal tumor, B) if the treatment is palliative in the metastatic setting, no additional requirements for tumor size or nodal involvement is needed; C) if the treatment is in the neoadjuvant setting, the tumor must ALSO be high-risk locally advanced rectal cancer defined as T3-4, N+, and/or at risk for a positive radial margin (as determined by the surgeon)
* For dose expansion: Patients must have A) histologically or cytologically confirmed rectal adenocarcinoma eligible for radiation therapy to rectal tumor irrespective of location from anal verge, B) if the treatment is palliative in the metastatic setting, no additional requirements for tumor size or nodal involvement is needed; C) if the treatment is in the neoadjuvant setting, the tumor must ALSO be high-risk locally advanced rectal cancer defined as T3-4, N+, and/or at risk for a positive radial margin (as determined by the surgeon)
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of talimogene laherparepvec in combination with chemotherapy in patients < 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000 x 10^9 /L
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert's syndrome, who can have total bilirubin < 3 mg/DL)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional unless the subject is on anticoagulant therapy (if the subject is receiving anticoagulant therapy, PT, and activated partial thromboplastin time [aPTT] must be within therapeutic range of intended use of anticoagulants)
* Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary; patients must be made aware of their other treatment options
* Talimogene laherparepvec, as well as other therapeutic agents used in this trial including radiation and capecitabine, may cause fetal harm when administered to a pregnant woman; women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; WOCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of the drug; WOCBP must have a negative serum pregnancy test within 72 hours prior to enrollment and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had radiotherapy within < 4 weeks are ineligible
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) except alopecia are ineligible
* Use of other investigational, chemotherapeutic or targeted drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of talimogene laherparepvec and during the study are ineligible
* Patients who have previously been treated with talimogene laherparepvec, any other oncolytic virus or pelvic radiation are ineligible
* Patients with known active central nervous system (CNS) metastases are ineligible; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases
* Patients with a known immediate or delayed hypersensitivity reaction or idiosyncrasy to talimogene laherparepvec or any of its components, capecitabine, fluorouracil (5-FU) and / or oxaliplatin are ineligible
* Patients with a history or evidence of active autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other); or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) within 2 months of enrollment are ineligible; (replacement therapy [e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency] is not considered a form of systemic treatment for autoimmune disease)
* Patients with evidence of clinically significant immunosuppression such as the following are ineligible:

  * Primary immunodeficiency state such as severe combined immunodeficiency disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
* Patients with active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis) are ineligible
* Patients with viral infections requiring intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use are ineligible
* Patients with other viral infections are ineligible:

  * Known to have acute or chronic active hepatitis B or hepatitis C infection
  * Known to have human immunodeficiency virus (HIV) infection
  * Prior therapy with viral-based tumor vaccine
  * Received live vaccine within 28 days prior to enrollment
* Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for herpes simplex virus (HSV)-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or children under the age of 1 year, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, active, non-colorectal malignancies requiring systemic therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are ineligible
* Although no effects on embryo-fetal development have been observed in animal studies, adequate and well-controlled studies with talimogene laherparepvec have not been conducted in pregnant women; in addition, given the high risk of detrimental effects of other study agents including capecitabine, 5-FU, oxaliplatin and radiation on embryo-fetal development, the study treatment must be excluded in the following patients:

  * Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 4 months after the last dose of talimogene laherparepvec
  * Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 4 months after the last dose of talimogene laherparepvec
  * Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec
* Patients that are unable to swallow oral medications are ineligible
* Patients with a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of therapy, or anticipation of need for major surgical procedure during the course of the study other than that defined by protocol are ineligible
* If patients require anticoagulation while on protocol, they should be switched from warfarin to another alternative anticoagulant such as low molecular weight heparin or oral direct factor Xa inhibitors as deemed appropriate by the treating physician for the duration they are on capecitabine (must be switched at least 1 week prior to starting capecitabine) to avoid drug-drug interaction of warfarin with capecitabine
* Patients with a known dihydropyrimidine dehydrogenase (DPD) deficiency are ineligible
* Patients who are unable to get MRIs due to any reason including pacemakers or automatic implantable cardioverter-defibrillator (AICD) are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwara V Dasari, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Talimogene Laherparepvec + FOLFOX + Short Course RT: Talimogene laherparepvec + FOLFOX + Short Course RT
Period: Overall Study
Arm/Group | Talimogene Laherparepvec + FOLFOX + Short Course RT
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Talimogene Laherparepvec + FOLFOX + Short Course RT (Radiation Therapy): Talimogene laherparepvec + FOLFOX + Short Course RT (Radiation Therapy)
Arm/Group | Talimogene Laherparepvec + FOLFOX + Short Course RT (Radiation Therapy)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Determination of Dose Limiting Toxicities (DLTs) and Maximum Tolerated Dose (MTD) of Talimogene Laherparepvec in Combination With Chemotherapy and Radiation in Rectal Cancer.
Description: Assessed using the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0.
Time Frame: 4 weeks after surgery
Population: Poor enrollment due to COVID-19 and change in standard of care led to discontinuation of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (T-VEC, Capecitabine, Chemoradiation)
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: To Establish Safety and Feasibility of the Combination
Description: Feasibility will be reported in all patients who have started therapy as percent of planned dose intensity. The scale for dose intensity will range from 0 - 100% with a higher score being better.
  The result will be reported using descriptive statistics.
Time Frame: 4 weeks after surgery
Population: Poor enrollment due to COVID-19 and change in standard of care led to discontinuation of the study
Measure: Median (Full Range); unit: percentage of dose intensity
Arm/Group | Treatment (T-VEC, Capecitabine, Chemoradiation)
Number analyzed (Participants) | 3
percentage of dose intensity | 99.5 [99 to 100]

3. Secondary Outcome: Determine the Neoadjuvant Rectal (NAR) Score of Talimogene Laherparepvec With Chemotherapy and Radiation.
Description: The NAR score has been validated in clinical trials as a surrogate endpoint for overall survival. The score is designed to be particularly sensitive to changes in factors that are affected by neoadjuvant. NAR is calculated based on the clinical T stage (cT), pathological T (pT) and pN stages as:
  NAR = [5pN- 3 (cT- pT) + 12] ^2 / 9.61 and will be reported using descriptive statistics
  Scale: The NAR score is a pseudo-continuous variable with 24 possible discrete scores from 0 to 100 with higher scores representing a poorer prognosis.
Time Frame: 4 weeks after surgery
Population: Poor enrollment due to COVID-19 and change in standard of care led to discontinuation of the study
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (T-VEC, Capecitabine, Chemoradiation)
Number analyzed (Participants) | 3
units on a scale | 30.07 [0.93 to 37.56]

ADVERSE EVENTS:
Time Frame: Baseline up to 12 weeks
Description: Poor enrollment due to COVID and change in standard of care led to discontinuation of the study.
Arm/Group | Treatment (T-VEC, Capecitabine, Chemoradiation)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (T-VEC, Capecitabine, Chemoradiation) (N=3)
Urinary frequency (Renal and urinary disorders) | 1
Pain (lower back) (Musculoskeletal and connective tissue disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Anemia (Investigations) | 1
ANC low (Investigations) | 2
Platelet count low (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Nervous system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03300544/Prot_SAP_000.pdf